CLINICAL TRIAL: NCT03743987
Title: Assessment of Bone Healing After MTA and PRF Application in Periapical Lesions By Using CBCT
Brief Title: The Effect of MTA and PRF Application in Periapical Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Nazife Begüm KARAN, Assistant Professor, DDS, PhD, Recep Tayyip Erdogan University Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RTEU 107
Record Dates: First submitted 2018-11-14; First posted 2018-11-16 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Apical Periodontitis; Wound Heal
MeSH Terms: conditions — Periapical Periodontitis | interventions — Control Groups; Apicoectomy; mineral trioxide aggregate; Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- control group (Sham Comparator): Apical resection group. Only root resection was applied without any other interventions (like prf or mta)
  Interventions: Procedure: control group
- MTA group (Experimental): Root resection was applied and MTA was inserted through the apical foramen
  Interventions: Procedure: MTA group
- PRF group (Experimental): Root resection was applied and PRF was placed to the surgically prepared area
  Interventions: Procedure: PRF group
- MTA + PRF group (Experimental): Root resection was applied. MTA was inserted through the apical foramen and PRF was placed to the surgically prepared area
  Interventions: Procedure: MTA + PRF group

INTERVENTIONS:
Procedure: control group — a procedure used to prevent or resolves apical periodontitis.
  Other Names: root resection
  Arms: control group
Procedure: MTA group — a procedure used to prevent or resolves apical periodontitis.
  Other Names: mineral trioxide aggregate
  Arms: MTA group
Procedure: PRF group — a procedure that is used for wound healing
  Other Names: platelet rich fibrin
  Arms: PRF group
Procedure: MTA + PRF group — a procedure used to prevent or resolves apical periodontitis in combination with a procedure that is used for wound healing.
  Other Names: mineral trioxide aggregate + mineral trioxide aggregate
  Arms: MTA + PRF group

SUMMARY:
A total of 40 periapical lesions from the 33 patient undergoing apical surgery were randomly selected from December 2016-November 2017. Patients were informed about the surgical procedure and signed a consent form. Groups were divided in to 4; as control, MTA (mineral trioxide aggregate), PRF (platelet rich fibrin) and MTA+PRF groups. Apical resection was performed in all groups. No other interventions were made to the control group.

Routine radiographs were taken in the 1st. 3th and 6th months. In the (approximately) 12th month of the procedures computerized tomography scans were taken. Primary healing of the periapical tissues were evaluated and the outcomes were measured. Patients have still been under control for the long term outcomes of the study.

DETAILED DESCRIPTION:
44 apically infected periapical lesions were decided to enroll to the study from December 2016-November 2017. However; a total of 40 periapical lesions undergoing apical surgery were recruited for the planned clinical trial in the end. The study was conducted under randomized controlled protocol. Patients were informed about the surgical procedures and signed a consent form. The anticipated outcomes, possible risks and benefits of the study as well as the alternative treatment options were explained to the patients.

Groups were designed to have 10 patients in each and randomly divided into four as; control, MTA, PRF and MTA+PRF. Apical resection was performed in all groups. No other interventions were made to the control group.

Routine radiographs were taken in the 1st. 3th and 6th months. In the 12th month of the procedures computerized tomography (CT) scans were taken. Primary healing of the periapical tissues were evaluated according to the volumes and the densities of the lesions. Outcomes were measured. Comparison between the initial and the last 3D CT scan volumes were made by medical image processing software (MIMICS, Belgium). Patients have still been under control for the long term outcomes of the study.

ELIGIBILITY:
Inclusion Criteria:

* Single rooted canals
* Failed previous root canal treatment
* Retreatment at least 1 year previously
* Previous surgery with unresolved bony lesion

Exclusion Criteria:

* More than single rooted canals
* Chronic generalized periodontitis
* Any systemic disease contraindicating oral surgical procedures
* Evidence of root fracture
* Resorptive processes involving more than apical third of the root

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2018-11-05 (Actual)

PRIMARY OUTCOMES:
Radiographic success - in volume | 1 year
  Evaluation of tomographic outcomes (differences between preoperative and postoperative volume of periapical lesions)
Radiographic success - in density | 1 year
  Evaluation of tomographic outcomes (differences between preoperative and postoperative density of periapical lesions)

CONTACTS AND LOCATIONS:
Overall Officials: Nazife Begüm KARAN, PhD, DDS, Principal Investigator — Recep Tayyip Erdogan University; Banu Arıcıoğlu, PhD, DDS, Principal Investigator — Recep Tayyip Erdogan University
Locations (1):
- Nazife Begüm KARAN, Ankara, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
data can be available 6 months after the acceptance of the paper

REFERENCES:
- [Derived] Karan NB, Aricioglu B. Assessment of bone healing after mineral trioxide aggregate and platelet-rich fibrin application in periapical lesions using cone-beam computed tomographic imaging. Clin Oral Investig. 2020 Feb;24(2):1065-1072. doi: 10.1007/s00784-019-03003-x. Epub 2019 Jul 18. PMID 31321573